CLINICAL TRIAL: NCT07099573
Title: Analysis of Hyperthermia as an Adjunctive Treatment to Evidence-based Clinical Intervention in Subjects With Bursitis: a Double-blind Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Manuel González-Sánchez, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 140/2025
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Bursitis; Hyperthermia
MeSH Terms: conditions — Bursitis; Hyperthermia | interventions — Diathermy; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hyperthermia 2 times per week (Experimental)
  Interventions: Radiation: Hyperthermia; Other: Physical Exercise; Other: Stretching
- Hyperthermia 3 times per week (Experimental)
  Interventions: Radiation: Hyperthermia; Other: Physical Exercise; Other: Stretching
- Non-Hyperthermia 2 times per week (Experimental)
  Interventions: Other: Physical Exercise; Other: Stretching
- Non-Hyperthermia 3 times per week (Experimental)
  Interventions: Other: Physical Exercise; Other: Stretching

INTERVENTIONS:
Radiation: Hyperthermia — Hyperthermia will be applied for a period of 15 to 20 minutes in the area to be treated, maintaining a thermal sensation of gentle heat for the patient and accompanied by active-assisted or passive mobilization of the structures adjacent to the bursa.
  Arms: Hyperthermia 2 times per week; Hyperthermia 3 times per week
Other: Physical Exercise — The therapeutic physical exercise will consist of 3 periods of isometric contraction of 30 seconds, with a rest period of 1 minute, varying the number of repetitions from 3 to 5 depending on the patient's symptoms.
Other: Stretching — Stretching of the involved muscles will involve 3 periods of maximum tolerable stretching without pain, lasting 20 seconds and resting for 30 seconds.

SUMMARY:
This project aims to analyze the use of hyperthermia within a bursitis treatment protocol, as well as to determine the difference between two and three sessions per week. Study participants will be divided into four intervention groups: the first will receive two sessions per week for a period of six months, while the second will receive three sessions per week for the same period. The treatment protocol will consist of therapeutic physical exercise focused on the affected joint, stretching of the involved muscles, and the application of hyperthermia to the bursa and surrounding areas. The third and fourth intervention groups will receive the same treatment as mentioned above, but without hyperthermia. The third group will receive three sessions per week, while the second group will receive two sessions per week. Two different types of measurement variables will be used: on the one hand, the objective variable will be measurement and assessment of the bursa using ultrasound imaging. Subjective measurement variables will also be used through validated questionnaires, which will address physical activity, perceived functional limitations, and the visual analog scale for pain perception.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis confirmed by performing an imaging test of Bursitis
* Have not yet received physiotherapy treatment.

Exclusion Criteria:

* Have undergone surgery.
* Those who refuse to participate in this study.
* Patients with muscle atrophy.
* Medical conditions that are contraindications for hyperthermia therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
DISABILITIES OF THE ARM, SHOULDER AND HAND QUESTIONNAIRE (DASH) | Baseline and up to one year
  It consists of a self-administered questionnaire that assesses the upper limb as a functional unit and allows for the quantification and comparison of the impact of different processes affecting different regions of the limb. It consists of a core of 30 items and two optional modules, each with four items. Each item is scored from 1 to 5, with higher scores corresponding to greater symptom intensity. The final score can range from 30 to 150 points, with a scale of 0 (best possible score) to 100 (worst possible score). The optional modules are scored separately. The Spanish version has very high reliability (r=0.96).
LOWER EXTREMITY FUNCTIONAL SCALE (LEFS) | This questionnaire assesses perceived functionality in patients with a musculoskeletal problem in the lower limb. It consists of 20 questions, each of which is scored by the patient, ranging from 0 (extreme difficulty or inability to perform the activity
International Physical Activity Questionnaire (IPAQ) | Baseline and up to one year
  This instrument is designed to measure physical activity levels in an adult population and can serve as a reference for making recommendations regarding physical activity. It comes in two versions: the long version with 31 items (IPAQ-LF) and the short version with 9 items (IPAQ-SF). The short version, which will be used in this study as recommended by the authors, measures activity at four intensity levels, ranging from 1 (vigorous-intensity activity) to 4 (sedentary). It has very good reliability (r=0.8).
Visual Analogue Scale (VAS) | Baseline and up to one year
  It consists of an 11-point numerical scale, ranging from 0 (no pain) to 10 (maximum pain intensity), which serves as a quantification for measuring pain intensity. It has moderate to good reliability.
Ultrasonography | Baseline and up to one year
  Ultrasound imaging techniques allow visualization of the bursa area, as the ultrasound beam can penetrate this region. These images enable detailed, multidimensional visualization of the joints and adjacent structures. They also allow precise differentiation of different tissue types, such as soft tissue, bone, or fluids. This is a noninvasive test; it involves placing the transducer on the skin surface, perpendicular to the anatomical location of the bursa.